CLINICAL TRIAL: NCT02472691
Title: Phase-II Trial to Assess the Efficacy and Safety of Lenalidomide in Addition to 5-Azacitidine and Donor Lymphocyte Infusions (DLI) for the Treatment of Patients With MDS, CMML or AML Who Relapse After Allogeneic Stem Cell Transplantation
Brief Title: Azacitidine, Lenalidomide and DLI as Salvage Therapy for MDS, CMML and sAML Relapsing After Allo-HSCT
Acronym: AZALENA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AZALENA-2013/RV-MDS-PI-0777
Record Dates: First submitted 2015-05-20; First posted 2015-06-16 (Estimated); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic
Keywords: relapse after allogeneic transplantation; MDS; AML; CMML; DLI; Azacitidine; Lenalidomide; C04.557.337.539.275; C15.378.190.625; C04.557.337.539.522
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic | interventions — Lenalidomide; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lenalidomide + Aza + DLI (Experimental): Patients will be included at the time of relapse after first allo-SCT. As standard of care all patients will receive Azacitidine 75 mg/m2/d for 7 days every 28 days for up to 8 cycles and DLIs given after cycle 4, 6 and 8 at a dose of 0.5-1x106CD3/kg (1st DLI), 1-5x106CD3/kg (2nd DLI) and 5-15x106CD3/kg (3rd DLI). As intervention (investigational drug), Lenalidomide will be also started on day 1 for 21 days every 28 days for a maximum of 8 cycles. Starting dose of Lenalidomide 2.5 mg per day for the first 10 patients. If no dose limiting toxicity is identified in a first interim analysis, the next 10 patients will be treated with 5 mg per day. In case of no DLT after a second interim analysis, the remaining 30 patients are envisaged to be treated with 5 mg per day.
  Interventions: Drug: Lenalidomide; Drug: Azacitidine; Biological: Donor Lymphocyte Infusions

INTERVENTIONS:
Drug: Lenalidomide — Lenalidomide (investigational drug) will be added to standard of care (Aza and DLI) starting from day 1 for 21 days every 28 days for a maximum of 8 cycles. Starting dose of Lenalidomide 2.5 mg per day for the first 10 patients. If no dose limiting toxicity is identified in a first interim analysis, the next 10 patients will be treated with 5 mg per day. In case of no DLT after a second interim analysis, the remaining 30 patients are envisaged to be treated with 5 mg per day.
  Other Names: Revlimid
Drug: Azacitidine — Starting on day 1 all patients will receive Azacitidine (standard of care) 75 mg/m2/d for 7 days every 28 days for up to 8 cycles.
  Other Names: Vidaza
Biological: Donor Lymphocyte Infusions — DLIs will be given after cycle 4, 6 and 8 at a dose of 0.5-1x10^6 CD3/kg (1st DLI), 1-5x10^6 CD3/kg (2nd DLI) and 5-15x10^6 CD3/kg (3rd DLI).
  Other Names: DLI

SUMMARY:
This is a prospective, open-label, single-arm multi-center phase II study aiming to evaluate the safety and feasibility of the addition of Lenalidomide (investigational drug) to the standard therapy of Azacitidine and DLI (standard of care) as first salvage therapy for relapse of MDS, CMML and AML with MDS-related changes (sAML, with 20%-30% bone marrow blasts, formerly RAEB-T) after allo-SCT. The starting dose of Lenalidomid is 2.5 mg per day for 21 days with a 7 day rest. The study incorporates 2 interim safety analyses after 10 and 20 patients in order to find the optimal and safe dose of Lenalidomide.

DETAILED DESCRIPTION:
This is a prospective, open-label, single-arm multi-center phase II study aiming to evaluate the safety and feasibility of the addition of Lenalidomide (investigational drug) to the standard therapy of Azacitidine and DLI (standard of care) as first salvage therapy for relapse of MDS, CMML and AML with MDS-related changes (sAML, with 20%-30% bone marrow blasts, formerly RAEB-T) after allo-SCT.

Study Design:

* prospective, open-label, single arm, multicenter phase-II trial
* total patients sample size: 50 patients
* number of trial sites: 6 all located in Germany and members of the EBMT Patients will be included at the time of relapse after first allo-SCT. Starting on day 1 all patients will receive Azacitidine 75 mg/m2/d for 7 days every 28 days for up to 8 cycles. DLIs will be given after cycle 4, 6 and 8. Lenalidomide will be also started on day 1 for 21 days every 28 days for a maximum of 8 cycles. The concomitant administration of Aza and Lenalidomide will be used since safety and efficacy of this schedule has been demonstrated.

Azacitidine and DLI represent a standard of care in this setting and are therefore not considered as investigational. As 5-Azacytidine is given in-label, treatment may be continued beyond 8 cycles. Additional DLIs may be given according to the investigators choice. However, to avoid severe GvHD it is recommended to give at least one more cycle 5-Azacytidine after additional DLIs.

The study incorporates a dose escalating schedule for Lenalidomide and two safety interim analyses. A first interim analysis will be performed as soon as 10 patients have been treated with Lenalidomide at a dose of 2.5mg/day If no dose limiting toxicity is observed in this cohort the next cohort of 10 patients will be treated with 5 mg per day for 21 days starting on day 1. If dose limiting toxicity occurs the study will be closed. A second interim analysis will be performed as soon as 10 patients have been treated with Lenalidomide at a dose of 5mg/day and the 10th patient of this cohort has either completed 4 cycles or has discontinued treatment whichever occurs first. If no dose limiting toxicity is observed in this cohort, the dose of 5 mg per day for 21 days starting on day 1 will be chosen and the remaining patients will be treated with this dose of Lenalidomide. If dose limiting toxicity occurs in patients treated with 5mg per day the remaining patients will be treated with Lenalidomide at a dose of 2.5mg/day. A total number of 50 patients will be treated.

Independent of the dose level, Lenalidomide will be stopped individually in the case of GvHD ≥ grade II.

ELIGIBILITY:
Inclusion Criteria:

* First relapse of de novo or therapy-related MDS, CMML or AML according to WHO classification (revised version 2016) without FLT3 mutation and without known IDH mutation after first allo-SCT (related or unrelated donor with < 2 HLA mismatches)
* Possibility of DLI (no cord blood, no haploidentical donor)
* no previous therapy for relapse after allo-SCT
* ECOG performance status ≤ 2 at study entry
* no active GvHD treated with systemic immunosuppression within 4 weeks before inclusion
* no uncontrolled infection at inclusion
* Understand and voluntarily sign an informed consent form.
* Age 18 years at the time of signing the informed consent form.
* Able to adhere to the study visit schedule and other protocol requirements.
* All females must acknowledge to have understood the hazards and necessary precautions associated with the use of lenalidomide

Exclusion Criteria:

* Relapse after second allogeneic Transplantation
* AML with FLT3 mutation (ITD or TKD)
* AML with known IDH mutation (IDH1 or IDH2)
* Any previous therapy (chemotherapy, radiation or investigational drugs) administered as therapy for relapse after allo-SCT
* previous transplantation with cord blood, an haploidentical donor or a related/unrelated donor with

  ≥2 HLA mismatches
* Active GvHD requiring systemic immunosuppression within the last 4 weeks
* Uncontrolled infection
* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
* Pregnant or lactating females
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study
* Impaired renal function (GFR < 20 ml/min)
* Impaired hepatic function
* Known hypersensitivity to thalidomide, lenalidomide or any components of the treatment
* The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
* Concurrent use of other anti-cancer agents or treatments.
* Known positive for HIV or infectious hepatitis, type A, B or C.
* Neuropathy ≥ grade 2
* Prior history of malignancy other than MDS or AML (except basal cell or squamous cell carcinoma or carcinoma in situ of the cervix or breast) unless the subject has been free of disease for ≥ 3 years
* Participation in another study with ongoing use of unlicensed investigational product from 28 days before study enrollment until the end of the study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2020-04-23 (Actual); Study Completion 2020-04-23 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety | 56 months (final analysis, two interim analysis after 10 and 20 patients)
  incidence and severity of adverse events
Type of Adverse Events as a Measure of Safety | 56 months (final analysis, two interim analysis after 10 and 20 patients)
  Type of adverse events
Severity of Adverse Events as a Measure of Safety | 56 months (final analysis, two interim analysis after 10 and 20 patients)
  Severity of Adverse Events

SECONDARY OUTCOMES:
Number of participants with responses according to International Working Group (IWG) criteria as a measure of efficacy | 8 months
  Best response within the first 8 months of treatment according to the International Working Group (IWG) criteria
Days from the beginning of treatment to best response in individual patients as a measure of efficacy | 56 months
  Time to response
Number of participants achieving complete donor chimerism as a measure of efficacy | 56 months
  Rate of complete donor chimerism
Number of participants with molecular response determined by disease-specific marker (e.g. FISH, mutations like TET2, ASXL1 etc.) or WT1 mRNA expression as a measure of efficacy | 56 months
  Molecular response measured by disease-specific marker (e.g. FISH, mutations like TET2, ASXL1 etc.) or WT1 mRNA expression
Days from beginning of remission to relapse as a measure of efficacy | 56 months
  Duration of remission
Days from start of treatment until death or last follow up as a measure of efficacy | 56 months
  Overall survival
Number of participants with a positive correlation between response and cytogenetics as a measure of efficacy | 56 months
  Correlation of response and cytogenetics/molecular alterations
Number of participants with acute GvHD according to Glucksberg Criteria as a measure of safety. | 56 months
  Incidence of aGvHD
Type of manifestations of acute GvHD according to Glucksberg Criteria as a measure of safety. | 56 months
  Type of aGvHD
Severity of acute GvHD manifestations according to Glucksberg Criteria as a measure of safety. | 56 months
  Severity of aGvHD
Number of hospitalizations per patients as a measure of safety | 56 months
  Number of hospitalizations
Number of participants with Adverse events specifying seriousness and expectedness (AE, SAE, SUSAR) according to ICH-GCP as a measure of safety. | 56 months
  Number of Adverse Events specifying seriousness and expectedness (AE, SAE, SUSAR)
Type of Adverse events specifying seriousness and expectedness (AE, SAE, SUSAR) according to ICH-GCP as a measure of safety. | 56 months
  Type of Adverse Events specifying seriousness and expectedness (AE, SAE, SUSAR)
Severity of Adverse events specifying seriousness and expectedness (AE, SAE, SUSAR) according to ICH-GCP as a measure of safety. | 56 months
  Severity of Adverse Events specifying seriousness and expectedness (AE, SAE, SUSAR)
Days from the beginning of treatment to complete donor chimerism as a measure of efficacy | 56 months
  Time to complete donor chimerisms
Number of participants with relapse as a measure of efficacy | 56 months
  Incidence of relapse
Number of participants with chronic GvHD according to NIH Consensus Criteria as a measure of safety. | 56 months
  Incidence of cGvHD
Type of manifestations of chronic GvHD according to NIH Consensus Criteria as a measure of safety. | 56 months
  Type of cGvHD
Severity of manifestations of chronic GvHD according to NIH Consensus Criteria as a measure of safety. | 56 months
  Severity of cGvHD

CONTACTS AND LOCATIONS:
Overall Officials: Guido Kobbe, Prof. Dr., Principal Investigator — University Hospital Duesseldorf, Dept. for Hematology, Oncology and Clinical Immunology
Locations (1):
- University Hospital Duesseldorf, Dept. of Hematology, Oncology and Clinical Immunology, Düsseldorf, North Rhine-Westphalia, Germany

REFERENCES:
- [Background] Schroeder T, Czibere A, Platzbecker U, Bug G, Uharek L, Luft T, Giagounidis A, Zohren F, Bruns I, Wolschke C, Rieger K, Fenk R, Germing U, Haas R, Kroger N, Kobbe G. Azacitidine and donor lymphocyte infusions as first salvage therapy for relapse of AML or MDS after allogeneic stem cell transplantation. Leukemia. 2013 Jun;27(6):1229-35. doi: 10.1038/leu.2013.7. Epub 2013 Jan 14. PMID 23314834
- [Result] Schroeder T, Rachlis E, Bug G, Stelljes M, Klein S, Steckel NK, Wolf D, Ringhoffer M, Czibere A, Nachtkamp K, Dienst A, Kondakci M, Stadler M, Platzbecker U, Uharek L, Luft T, Fenk R, Germing U, Bornhauser M, Kroger N, Beelen DW, Haas R, Kobbe G. Treatment of acute myeloid leukemia or myelodysplastic syndrome relapse after allogeneic stem cell transplantation with azacitidine and donor lymphocyte infusions--a retrospective multicenter analysis from the German Cooperative Transplant Study Group. Biol Blood Marrow Transplant. 2015 Apr;21(4):653-60. doi: 10.1016/j.bbmt.2014.12.016. Epub 2014 Dec 23. PMID 25540937
- [Derived] Schroeder T, Stelljes M, Christopeit M, Esseling E, Scheid C, Mikesch JH, Rautenberg C, Jager P, Cadeddu RP, Drusenheimer N, Holtick U, Klein S, Trenschel R, Haas R, Germing U, Kroger N, Kobbe G. Azacitidine, lenalidomide and donor lymphocyte infusions for relapse of myelodysplastic syndrome, acute myeloid leukemia and chronic myelomonocytic leukemia after allogeneic transplant: the Azalena-Trial. Haematologica. 2023 Nov 1;108(11):3001-3010. doi: 10.3324/haematol.2022.282570. PMID 37259567